CLINICAL TRIAL: NCT01400295
Title: Predictive Value of the Contrast Media Volume to Creatinine Clearance Ratio for the Risk of Contrast-Induced Nephropathy After Coronary Angiography
Brief Title: PREdictive Value of COntrast voluMe to creatinINe Clearance Ratio
Acronym: PRECOMIN
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Chen, MD, Guangdong Provincial People's Hospital
Other Study IDs: 20100917
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast-induced nephropathy; contrast medium; creatinine clearance; coronary angiography; diabetes; chronic kidney disease
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary angiography: The investigators reviewed all consecutive patients who were undergoing coronary angiography

SUMMARY:
To determine a relatively safe contrast media volume to creatinine clearance cut-off value to avoid contrast-induced nephropathy in patients following coronary angiography

DETAILED DESCRIPTION:
Contrast media volume to creatinine clearance (V/CrCl) ratios were obtained from consecutive consenting patients after coronary angiography. Receiver-operator characteristic (ROC) curves were used to identify the optimal sensitivity for the observed range of V/CrCl. The predictive value of V/CrCl for the risk of contrast-induced nephropathy was assessed using multivariate logistic regression.Subgroup analysis was performed on patients with creatinine clearance < 60 ml/min,diabetes,emergent angiography.

ELIGIBILITY:
Inclusion Criteria:

* patients who agreed to stay in the hospital for 2-3 days after coronary angiography
* provided written informed consent

Exclusion Criteria:

* pregnancy
* lactation
* intravascular administration of an contrast medium within the previous seven days
* treatment with metformin,aminoglycosides,N-acetylcysteine (NAC),nonsteroidal anti-inflammatory drugs within the previous 48 h
* intake of nephrotoxic drugs within the previous seven days
* history of serious reactions to contrast mediums， severe concomitant disease renal transplantation , or end-stage renal disease necessitating dialysis
* patients who died during coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators reviewed all consecutive patients who were undergoing coronary angiography
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Contrast-Induced Nephropathy | 48-72 h
  Contrast-Induced Nephropathy was defined as an increase in serum creatinine of more than 0.5 mg/dl from the baseline within 48-72 h of contrast exposure

SECONDARY OUTCOMES:
An early abnormal increase in serum creatinine | 24h
  An early abnormal increase in serum creatinine defined as an increase in serum creatinine of more than 0.5 mg/dl from the baseline within 24h of contrast exposure
Major adverse clinical events | 1 year
  Major adverse clinical events: death, requiring renal replacement therapy, 2nd myocardial infarction,target revascularization,acute heart failure, mechanical ventilation,2nd angina,tachyarrhythmia,hypotension,intra-aortic balloon pump and stroke
Major adverse clinical events | 1month
  Major adverse clinical events: death, requiring renal replacement therapy, 2nd myocardial infarction,target revascularization,acute heart failure, mechanical ventilation,2nd angina,tachyarrhythmia,hypotension,intra-aortic balloon pump and stroke
An early abnormal increase in serum cystatin C | 24h
  An early abnormal increase in serum cystatin C was defined as an increase more than 10% from the baseline within 24h of contrast exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, MD, Study Chair — Guangdong Cardiovascular Institute,Guangdong General Hospital; Yong Liu, MD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Yingling Zhou, MD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Ning Tan, MD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Jianfang Luo, MD, Principal Investigator — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (1):
- Guangdong Cardiovascular Institute,Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu L, Liu J, Lei L, Wang B, Sun G, Guo Z, He Y, Song F, Lun Z, Liu B, Chen G, Chen S, Yang Y, Liu Y, Chen J. A prediction model of contrast-associated acute kidney injury in patients with hypoalbuminemia undergoing coronary angiography. BMC Cardiovasc Disord. 2020 Aug 31;20(1):399. doi: 10.1186/s12872-020-01689-6. PMID 32867690
- [Derived] Liu Y, Chen S, Ye J, Xian Y, Wang X, Xuan J, Tan N, Li Q, Chen J, Ni Z. Random forest for prediction of contrast-induced nephropathy following coronary angiography. Int J Cardiovasc Imaging. 2020 Jun;36(6):983-991. doi: 10.1007/s10554-019-01730-6. Epub 2020 Apr 13. PMID 32285318
- [Derived] Liu J, Sun G, He Y, Song F, Chen S, Guo Z, Liu B, Lei L, He L, Chen J, Tan N, Liu Y. Early beta-blockers administration might be associated with a reduced risk of contrast-induced acute kidney injury in patients with acute myocardial infarction. J Thorac Dis. 2019 Apr;11(4):1589-1596. doi: 10.21037/jtd.2019.04.65. PMID 31179103
- [Derived] Guo XS, Chen SQ, Duan CY, Li HL, Bei WJ, Liu Y, Tan N, Chen PY, Chen JY. Association of post-procedural early (within 24h) increases in serum creatinine with all-cause mortality after coronary angiography. Clin Chim Acta. 2017 Nov;474:96-101. doi: 10.1016/j.cca.2017.08.036. Epub 2017 Sep 1. PMID 28866117